CLINICAL TRIAL: NCT02493413
Title: The Stress-release Effects of Exercise in Obese Are Determined by DS14 Score and T-cell Activation Status
Status: Completed | Type: Observational
Sponsor: Institute for Preventive Medicine, Trzaska (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Mateja Hafner M.D., M.D., Institute for Preventive Medicine, Trzaska
Other Study IDs: 001563777
Record Dates: First submitted 2015-07-01; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Obesity; Type D Personality; Coronary Heart Disease
Keywords: psychoneuroimmunology; stress; lymphocyte population; personality type; obesity; heart rate variability; awareness
MeSH Terms: conditions — Obesity; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: observational time of three months in the obese group with distressed (type D) personality (high DS 14 score) with moderate aerobic exercise
- Group B: observational time of three months in obese group without distressed personality (low DS 14 score) with moderate aerobic exercise

SUMMARY:
The purpose of the study was to analyze negative affectivity (NA) and social inhibition (SI) inquired by DS14 score in type D personality (distressed personality) to the relation of autonomic regulation of heart function (HRV) and immune response (T lymphocyte) among obese patients within coronary heart disease group (CHD). As stress is the key psychological activator of the hypothalamic-pituitary-adrenal axis (HPA axis) and therefore an important risk factor for diminished immune competency and prevalence of chronic conditions such as obesity, investigators chose exercise as the stress release intervention, especially as chronic stress may have a role in obesity, related to initiation or exacerbation of the condition. Abnormal regulation of the hypothalamic-pituitary-adrenal axis is additionally associated with chronic inflammatory conditions. Proinflammatory T-lymphocytes are present in visceral adipose tissue and may contribute to local inflammatory cell activation before the appearance of macrophages, suggesting that these cells could play an important role in the initiation and perpetuation of adipose tissue inflammation.

DETAILED DESCRIPTION:
This study was performed at The Institute for Preventive Medicine in cooperation with The Institute of Microbiology and Immunology at the Medical Faculty of Ljubljana/University of Ljubljana in a clinical setting as an observational type. In the group of examinees the investigators chose only those obese without detectable complications of coronary heart disease while admitted. Obese patients with angina pectoris, myocardial infarction, valvular heart disease and congestive heart disease had been excluded from the research. Since personality is the major determinant of chronic stress, according to the investigators hypothesis, further division on two global traits Negative affectivity (NA) and Social inhibition (SI) structured by Denollet has been positioned in the study. A total of 30 patients with CHD were divided in two groups. Participants who were obese with high DS14 score matched obese controls with normal DS14 score. In all subjects the investigators also observed white blood cell counts with a detailed lymphocyte analysis using flow cytometry and C-reactive protein (CRP) as the indicator of inflammation. Besides body mass (BM), body mass index (BMI) systolic and diastolic blood pressure (SBP, DBP), heart rate (HR), and heart rate variability (HRV) were measured before and after three months period, while all subjects had been already exercising 4 times weakly (moderate walking of 5km/h) for an hour. Additionally STAIX-1, SWLS and QOLLTI-P questionnaires had been used.

ELIGIBILITY:
Inclusion Criteria:

* obese people without detectable complications of coronary heart disease

Exclusion Criteria:

* Obese patients with angina pectoris, myocardial infarction, valvular heart disease and congestive heart disease had been excluded from the research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 examinees, 14 men of average age 56,3 ± 15,5 years old and 16 women of average age of 53,5. ± 4,2 years old made the owerweight/obese group of chronic (coronary heart disease) patients. Subjects were matched by gender, age, body mass index and had all been regular visitors (patients) of The Institute of Preventive Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in DS14 Score at 3 Months | baseline and 3 months
  Each examines filled in DS14 scale to determine negative affectivity (NA), social inhibition (SI) and Type D personality for early identification of high-risk CHD patients (Denollet, 2005). Subjects rated their personality on a 5-point Likert scale ranging from 0 _ false to 4 _true. The NA and SI scales can be scored as continuous variables (range, 0-28) to assess these personality traits in their own right. A cutoff of 10 on both scales is used to classify subjects as Type D (NA _10 and SI _10).
Change in STAIX-1 questionnaire score | baseline and 3 months
  The STAIX-1 Form is an administered analysis of reported anxiety symptoms. The first subscale measures state anxiety, the second measures trait anxiety.
  The range of scores is 20-80, the higher the score indicating greater anxiety.
Change in Peripheral Human Blood Leucocytes | baseline and 3 months
  Peripheral human blood leucocytes were collected by the venipuncture procedure and collected into Vacutainers.Two-parameter analysis was performed to determine the proportion of T cells (CD3+), T helper cells (CD3+CD4+) and cytotoxic T cells (CD3+CD8+). Isotype controls (Becton Dickinson, Mountain View, CA) and a control of viable cells (LIVE/DEAD kit, Molecular Probes, OR) were included. At least 2000 gated cells were analyzed for each test, and signals from two light scatters and four fluorescence parameters were analyzed with the Becton Dickinson Lysis II software.
Change in Cortisol Levels | baseline and 3 months
  The measurement of cortisol in salivary samples accurately reflects levels of physiologically active unbound (free) cortisol in the blood, which diffuses from the blood to saliva.
Change in Heart Rate variability (HRV) | baseline and 3 months
  The investigators chose the combination of Time domain methods and Frequency domain methods to compare variability among groups under physical exercise and within 24 hours.
Change in SWLS questionnaire score | baseline and 3 months
  The Satisfaction With Life Scale (SWLS) is a measure of life satisfaction. Life satisfaction can be assessed specific to a particular domain of life (e.g., work, family) or globally. The SWLS is a global measure of life satisfaction.
Change in QOLLTI-P questionnaire score | baseline and 3 months
  The Quality of Life in Life-Threatening Illness-Patient questionnaire (QOLLTI-P) is a self-administered questionnaire based on the McGill Quality of Life questionnaire (MQOL) with domains added to enhance content validity. Participants were asked to complete a set of above questionnaires prior to immunological assessment and HRV measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Mateja Hafner, M.D., Principal Investigator — Institute of Preventive medicine

REFERENCES:
- [Background] Denollet J. DS14: standard assessment of negative affectivity, social inhibition, and Type D personality. Psychosom Med. 2005 Jan-Feb;67(1):89-97. doi: 10.1097/01.psy.0000149256.81953.49. PMID 15673629
- [Background] Suwa A, Shimokawa T. Emerging targets for the treatment of obesity. FEBS J. 2011 Feb;278(4):551. doi: 10.1111/j.1742-4658.2010.07981.x. Epub 2010 Dec 30. No abstract available. PMID 21291513
- [Background] Kintscher U, Hartge M, Hess K, Foryst-Ludwig A, Clemenz M, Wabitsch M, Fischer-Posovszky P, Barth TF, Dragun D, Skurk T, Hauner H, Bluher M, Unger T, Wolf AM, Knippschild U, Hombach V, Marx N. T-lymphocyte infiltration in visceral adipose tissue: a primary event in adipose tissue inflammation and the development of obesity-mediated insulin resistance. Arterioscler Thromb Vasc Biol. 2008 Jul;28(7):1304-10. doi: 10.1161/ATVBAHA.108.165100. Epub 2008 Apr 17. PMID 18420999
- [Background] Ader R, Cohen N. Behaviorally conditioned immunosuppression. Psychosom Med. 1975 Jul-Aug;37(4):333-40. doi: 10.1097/00006842-197507000-00007. PMID 1162023
- [Background] Thayer JF, Ahs F, Fredrikson M, Sollers JJ 3rd, Wager TD. A meta-analysis of heart rate variability and neuroimaging studies: implications for heart rate variability as a marker of stress and health. Neurosci Biobehav Rev. 2012 Feb;36(2):747-56. doi: 10.1016/j.neubiorev.2011.11.009. Epub 2011 Dec 8. PMID 22178086
- [Background] Watson D, Pennebaker JW. Health complaints, stress, and distress: exploring the central role of negative affectivity. Psychol Rev. 1989 Apr;96(2):234-54. doi: 10.1037/0033-295x.96.2.234. PMID 2710874
- [Background] Denollet J. Negative affectivity and repressive coping: pervasive influence on self-reported mood, health, and coronary-prone behavior. Psychosom Med. 1991 Sep-Oct;53(5):538-56. doi: 10.1097/00006842-199109000-00005. PMID 1758940
- [Background] Friedman HS, Booth-Kewley S. Personality, type A behavior, and coronary heart disease: the role of emotional expression. J Pers Soc Psychol. 1987 Oct;53(4):783-92. doi: 10.1037//0022-3514.53.4.783. PMID 3681651
- [Background] Gest SD. Behavioral inhibition: stability and associations with adaptation from childhood to early adulthood. J Pers Soc Psychol. 1997 Feb;72(2):467-75. doi: 10.1037//0022-3514.72.2.467. PMID 9107012
- [Background] Denollet J, Sys SU, Brutsaert DL. Personality and mortality after myocardial infarction. Psychosom Med. 1995 Nov-Dec;57(6):582-91. doi: 10.1097/00006842-199511000-00011. PMID 8600485
- [Background] Denollet J, Sys SU, Stroobant N, Rombouts H, Gillebert TC, Brutsaert DL. Personality as independent predictor of long-term mortality in patients with coronary heart disease. Lancet. 1996 Feb 17;347(8999):417-21. doi: 10.1016/s0140-6736(96)90007-0. PMID 8618481
- [Background] Ferguson E, Ward JW, Skatova A, Cassaday HJ, Bibby PA, Lawrence C. Health specific traits beyond the Five Factor Model, cognitive processes and trait expression: replies to Watson (2012), Matthews (2012) and Haslam, Jetten, Reynolds, and Reicher (2012). Health Psychol Rev. 2013 May;7(Suppl 1):S85-S103. doi: 10.1080/17437199.2012.701061. Epub 2013 May 28. PMID 23772232
- [Background] Piestrzeniewicz K, Luczak K, Lelonek M, Wranicz JK, Goch JH. Obesity and heart rate variability in men with myocardial infarction. Cardiol J. 2008;15(1):43-9. PMID 18651384
- [Background] Lee DC, Pate RR, Lavie CJ, Sui X, Church TS, Blair SN. Leisure-time running reduces all-cause and cardiovascular mortality risk. J Am Coll Cardiol. 2014 Aug 5;64(5):472-81. doi: 10.1016/j.jacc.2014.04.058. PMID 25082581
- [Background] Thayer JF, Sternberg E. Beyond heart rate variability: vagal regulation of allostatic systems. Ann N Y Acad Sci. 2006 Nov;1088:361-72. doi: 10.1196/annals.1366.014. PMID 17192580
- [Background] Hirsch JA, Bishop B. Respiratory sinus arrhythmia in humans: how breathing pattern modulates heart rate. Am J Physiol. 1981 Oct;241(4):H620-9. doi: 10.1152/ajpheart.1981.241.4.H620. PMID 7315987
- [Background] O'Keefe JH, Lavie CJ. Run for your life ... at a comfortable speed and not too far. Heart. 2013 Apr;99(8):516-9. doi: 10.1136/heartjnl-2012-302886. Epub 2012 Nov 29. No abstract available. PMID 23197444
- [Background] Malfatto G, Facchini M, Sala L, Branzi G, Bragato R, Leonetti G. Effects of cardiac rehabilitation and beta-blocker therapy on heart rate variability after first acute myocardial infarction. Am J Cardiol. 1998 Apr 1;81(7):834-40. doi: 10.1016/s0002-9149(98)00021-6. PMID 9555771
- [Background] Turnbull AV, Rivier C. Regulation of the HPA axis by cytokines. Brain Behav Immun. 1995 Dec;9(4):253-75. doi: 10.1006/brbi.1995.1026. PMID 8903845
- [Background] Yasuma F, Hayano J. Respiratory sinus arrhythmia: why does the heartbeat synchronize with respiratory rhythm? Chest. 2004 Feb;125(2):683-90. doi: 10.1378/chest.125.2.683. PMID 14769752
- [Background] Hrushesky WJ, Fader D, Schmitt O, Gilbertsen V. The respiratory sinus arrhythmia: a measure of cardiac age. Science. 1984 Jun 1;224(4652):1001-4. doi: 10.1126/science.6372092.
- [Background] Steptoe A, Brydon L. Emotional triggering of cardiac events. Neurosci Biobehav Rev. 2009 Feb;33(2):63-70. doi: 10.1016/j.neubiorev.2008.04.010. Epub 2008 May 3. PMID 18534677